CLINICAL TRIAL: NCT03457766
Title: Presurgical Evaluation of Nonmelanoma Skin Cancers Using High Frequency Ultrasound
Brief Title: Presurgical Evaluation of Skin Cancers Using HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, George Gamil Gergis, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HIFU in skin cancers
Record Dates: First submitted 2018-02-24; First posted 2018-03-08 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Skin Cancer, Non-Melanoma
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: Using high frequency ultrasound in identification of safety margins of skin cancers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with skin lesions (Experimental): Using HIFU in identification of safety margins of lesions clinically apparent locally malignant, or malignant
  Interventions: Device: HIFU

INTERVENTIONS:
Device: HIFU — Ultrasound (Esaota MyLabSeven) imaging system using (SL2325) probe with (6-19 MHz) frequency
  Other Names: Esaota MyLabSeven

SUMMARY:
1. To ensure complete elimination of lesions with maximum preservation of function and aesthetics.
2. To elaborate the Ultrasonographic features of skin cancers.
3. To determine the accuracy of HIFU to assess the margins of skin lesions and its safety margins by histopathiological examination..
4. To follow up the patient postoperatively for incomplete excision or recurrence by clinical and HIFU examination.

DETAILED DESCRIPTION:
The skin is the most superficial and largest body organ, due to its function as a surface covering for the body, enables the performance of noninvasive diagnostic and investigative procedures.

Of all the tumors that affect humans, non-melanoma cutaneous cancer is the most common e.g. basal cell carcinoma (BCC) and squamous cell carcinoma (SCC).

Techniques such as high frequency ultrasound (HFUS) enable the real-time study of cutaneous lesions, making them excellent pre-operative tools varying considerably in their penetration, resolution, and applicability.

High frequency ultrasound has been used in dermatology since the 1970s, ultrasonography is a painless non-radioactive imaging diagnostic method based on the reflection of sound waves through body tissues.

High frequency ultrasound allows for the delimiting of the margins of the neoplasia, due to the difference in echogenicity between the hypoechoic tumoral area and the hyperechoic perilesional area.

High frequency ultrasound examination of each lesion should consist of:

1. A morphologic study analyzing the structural sonographic pattern and margins;
2. the measurement of the largest transverse diameter and thickness;
3. Color Doppler USG for perilesional vessels ; and
4. in cases suspicious for malignancy, the surrounding areas are scanned for locoregional metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 30 & 80 years.
* Lesions clinically apparent locally malignant, or malignant.
* Lesions with or without visible ulcerations.

Exclusion Criteria:

* Surgeon unable to visualize tumor on clinical examination.
* Patients unfit for surgery.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Complete excision of nonmelanoma skin cancers | Baseline
  Determination the accuracy of HIFU to assess the margins of skin lesions and its safety margins to ensure complete elimination of lesions with maximum preservation of function and aesthetics

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa AH El-Sonbaty, Professor, Study Chair — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Proksch E, Brandner JM, Jensen JM. The skin: an indispensable barrier. Exp Dermatol. 2008 Dec;17(12):1063-72. doi: 10.1111/j.1600-0625.2008.00786.x. PMID 19043850
- [Background] Eggermont AM, Spatz A, Robert C. Cutaneous melanoma. Lancet. 2014 Mar 1;383(9919):816-27. doi: 10.1016/S0140-6736(13)60802-8. Epub 2013 Sep 19. PMID 24054424
- [Background] Madan V, Lear JT, Szeimies RM. Non-melanoma skin cancer. Lancet. 2010 Feb 20;375(9715):673-85. doi: 10.1016/S0140-6736(09)61196-X. PMID 20171403
- [Background] Kleinerman R, Whang TB, Bard RL, Marmur ES. Ultrasound in dermatology: principles and applications. J Am Acad Dermatol. 2012 Sep;67(3):478-87. doi: 10.1016/j.jaad.2011.12.016. Epub 2012 Jan 30. PMID 22285673
- [Background] Bobadilla F, Wortsman X, Munoz C, Segovia L, Espinoza M, Jemec GB. Pre-surgical high resolution ultrasound of facial basal cell carcinoma: correlation with histology. Cancer Imaging. 2008 Sep 22;8(1):163-72. doi: 10.1102/1470-7330.2008.0026. PMID 18812268
- [Background] Diepgen TL, Mahler V. The epidemiology of skin cancer. Br J Dermatol. 2002 Apr;146 Suppl 61:1-6. doi: 10.1046/j.1365-2133.146.s61.2.x. PMID 11966724
- [Background] Essers BA, Dirksen CD, Nieman FH, Smeets NW, Krekels GA, Prins MH, Neumann HA. Cost-effectiveness of Mohs Micrographic Surgery vs Surgical Excision for Basal Cell Carcinoma of the Face. Arch Dermatol. 2006 Feb;142(2):187-94. doi: 10.1001/archderm.142.2.187. PMID 16490846
- [Background] Ansarin H, Daliri M, Soltani-Arabshahi R. Expression of p53 in aggressive and non-aggressive histologic variants of basal cell carcinoma. Eur J Dermatol. 2006 Sep-Oct;16(5):543-7. PMID 17101476